CLINICAL TRIAL: NCT01575223
Title: The HVSI STUDY: High Volume Saline Irrigation in the Post-operative Management of Chronic Rhinosinusitis: A Multicenter Randomized Single-Blind Controlled Trial
Brief Title: Saline Irrigation After Surgery in Patients With Chronic Sinusitis
Acronym: HVSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: NeilMed Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Kristian Macdonald, Principal Investigator, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HVSI-001
Record Dates: First submitted 2012-04-01; First posted 2012-04-11 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Rhinosinusitis
Keywords: saline irrigation; chronic rhinosinusitis; endoscopic sinus surgery; high volume saline irrigation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume saline irrigation (Active Comparator): Patients in this group will receive high volume saline irrigation (NeilMed sinus rinse)
  Interventions: Device: NeilMed sinus rinse
- Placebo (Placebo Comparator): Patients in this group will receive low volume saline irrigation (Salinex)
  Interventions: Device: Salinex

INTERVENTIONS:
Device: NeilMed sinus rinse — High volume saline irrigation
  Arms: High volume saline irrigation
Device: Salinex — Low volume saline irrigation
  Arms: Placebo

SUMMARY:
Purpose: To determine if high volume saline nasal irrigation (HVSI), (NeilMed® Sinus Rinse™) offers a benefit over low volume saline irrigation (LVSI), (Salinex®) in the early post-operative management in patients with chronic rhino sinusitis.

DETAILED DESCRIPTION:
Background: Chronic Rhinosinusitis (CRS) is a common inflammatory condition of the upper respiratory tract lasting more than 8 to 12 weeks. Major symptoms include facial congestion/fullness, facial pain/pressure, nasal obstruction/blockage, purulent nasal drainage, and reduction or loss of smell. The diagnosis must include two major symptoms and either endoscopic evidence of polyps, edema or mucopurulent discharge from the middle meatus and/or CT changes in the mucosa of sinuses or osteomeatal complexes.1

CRS has an estimated prevalence of 5% in the Canadian population2, and up to 16% in some adult populations in the United States.3 Sinusitis is associated with a major societal health care burden, costing billions of dollars a year in North America.4,5 The medical treatment of CRS includes topical saline and corticosteroid sprays, systemic steroids and antimicrobials. Specifically, saline nasal irrigation (SNI) is a safe, nonpharmacologic treatment, and an important and efficacious component in the management of CRS.6,7 SNI can vary by concentration (e.g. hypertonic, isotonic, hypotonic) and device (e.g. bulb syringe, nasal mist, squeeze bottle).

The Mayo Clinic recently reviewed major expert consensus guidelines on the medical treatment of CRS.8 Although they recognized an overall paucity of controlled trials for any medical treatment, and a lack of a consensus or algorithm in the treatment of CRS, there is an overall consensus agreement of the use for SNI in this population. In this review, there was no mention of treatment of CRS in postoperative period, and no recommendation of what type of SNI is best.

Few studies examine various SNI formulations in the postoperative period. These were highlighted by Canadian authors in a recent exhaustive review of SNI in sinusitis.9 Three studies, all greater than 15 years old, include formulations that are not currently in popular use, or even available in North America.10-12 These did show that pressurized jets or sprays of seawater were more effective than nasal drops. More recently, Harvey et al. examined how irrigation is delivered and retained in the sinus, using more common devices.13,14 In a cadaveric model, they compared HVSI to LVSI devices and found a greater delivery (p<..02) in the former. To date there are no studies comparing HVSI to LVSI, using subjective patient benefit and objective endoscopic measure outcomes, in the postoperative CRS patient.

One study did examine two different SNI devices in the management of CRS.15 The authors recruited 150 subjects with CRS in the primary care setting, and randomized them to two weeks of SNI with a bulb syringe, SNI with a nasal irrigation pot, and a control group of reflexology massage.15 Hypertonic saline was used in both treatment groups. Subjective questionnaires were administered at baseline and at the end of the study period. Both groups significantly improved, with no significant difference between the two SNI devices. Patients equally preferred the two devices.

Popular HVSI and LVSI formulations with patients and physicians are NeilMed® Sinus Rinse™ and Salinex®, respectively. These are two examples of positive pressure treatments,13 which have enjoyed widespread usage in North America preceding sufficient evidence-based medicine demonstrating safety and efficacy. This is likely because topical saline sprays are considered safe; they do not require a prescription, and perhaps most importantly the massive marketing campaign surrounding SNI devices. SNI devices have received significant news coverage and appearances on major television shows, including the Oprah Winfrey Show, the New York Times, and numerous YouTube videos.16 Purpose: The authors hypothesize that there is an advantage of HVSI over LVSI. The mechanical effect of high volume irrigation helps ensure that a larger surface area of sinonasal mucosa is debrided and cleansed.

The aim of this study is to determine if there is a clinical benefit of HVSI over LVSI in the postoperative period in patients with CRS. This information would help otolaryngologists, family physicians, and other health care professionals recommend the best SNI device for their patients with CRS. It would also provide a much-needed prospective and controlled trial in the evidence for SNI in CRS in the post-operative period.

Population/Procedure: This is a multicenter, randomized, single blind, controlled prospective study evaluating the subjective and objective outcomes of HSVI versus LSVI in patients who have ESS for CRS. One month postoperative scores will be compared to preoperative scores. The expected total number of patients to be enrolled in this study is approximately 100, with a planned completion time of one year.

At our institution, ten patients who are offered endoscopic sinus surgery (ESS) for CRS will be approached for study participation.

ELIGIBILITY:
Inclusion criteria:

* Documented diagnosis of unilateral or bilateral CRS
* Documented failed medical treatment of CRS
* Eighteen (18) to sixty-five (65) years of age
* Planned ESS for the treatment of CRS
* Able to read and understand English

Exclusion criteria:

* Pregnant
* Cystic Fibrosis
* Diagnosed immotile cilia syndrome
* Diagnosed immunodeficiency syndrome
* Diagnosed fungal sinusitis
* Sinonasal tumours or obstructive lesions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Sinonasal Outcomes Scale (SNOT-22) | One month post-operatively
  Subjective scale, completed by patient. Validated scale for chronic sinusitis.
Lund MacKay score | 1 month postoperatively
  Objective scale, validated, completed by investigator. Preoperative CT scan is scored based on degree of sinus opacification (0-24).
Nasal and Sinus Symptom Score (NSS) - Subjective scale | 1 month post-operatively
  A subjective scale, filled out by the patient, specific to symptoms of sinusitis.
Perioperative Sinus Endoscopy scale (POSE) | 1 month post-operatively
  Objective scale, completed by treating physician, to assess sinonasal contents endoscopically. Validated scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Witterick, MD MSc FRCSC, Principal Investigator — Samuel R Lunenfeld Institute
Locations (4):
- Canada (4):
  - University of Calgary Otolaryngology - Head & Neck Surgery, Calgary, Alberta
  - Western University Dept. of Otolaryngology - Head & Neck Surgery, London, Ontario
  - Ottawa University Otolaryngology - Head & Neck Surgery, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Background] Desrosiers M, Evans GA, Keith PK, Wright ED, Kaplan A, Bouchard J, Ciavarella A, Doyle PW, Javer AR, Leith ES, Mukherji A, Robert Schellenberg R, Small P, Witterick IJ. Canadian clinical practice guidelines for acute and chronic rhinosinusitis. J Otolaryngol Head Neck Surg. 2011 May;40 Suppl 2:S99-193. English, French. PMID 21658337
- [Background] Chen Y, Dales R, Lin M. The epidemiology of chronic rhinosinusitis in Canadians. Laryngoscope. 2003 Jul;113(7):1199-205. doi: 10.1097/00005537-200307000-00016. PMID 12838019
- [Background] Anand VK. Epidemiology and economic impact of rhinosinusitis. Ann Otol Rhinol Laryngol Suppl. 2004 May;193:3-5. doi: 10.1177/00034894041130s502. PMID 15174752
- [Background] Ray NF, Baraniuk JN, Thamer M, Rinehart CS, Gergen PJ, Kaliner M, Josephs S, Pung YH. Healthcare expenditures for sinusitis in 1996: contributions of asthma, rhinitis, and other airway disorders. J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):408-14. doi: 10.1016/s0091-6749(99)70464-1. PMID 10069873
- [Background] Harvey RJ, Debnath N, Srubiski A, Bleier B, Schlosser RJ. Fluid residuals and drug exposure in nasal irrigation. Otolaryngol Head Neck Surg. 2009 Dec;141(6):757-61. doi: 10.1016/j.otohns.2009.09.006. PMID 19932850